CLINICAL TRIAL: NCT07278518
Title: CTN-0156: Pilot Development and Evaluation of a Patient Decision Aid for Emergency Department Initiated Buprenorphine
Brief Title: Evaluation of a Patient Decision Aid for Emergency Department Initiated Buprenorphine
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Lindsey Jennings, Associate Professor-Faculty, Medical University of South Carolina
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: Pro00145434
Record Dates: First submitted 2025-12-03; First posted 2025-12-12 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2025-08

CONDITIONS: Opioid Use Disorder
Keywords: buprenorphine; patient decision aid; emergency department
MeSH Terms: conditions — Opioid-Related Disorders; Emergencies

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patient Decision Aid (Experimental): This arm will receive the patient decision aid
  Interventions: Behavioral: Patient Decision Aid for Opioid Use Disorder
- Treatment as Usual (No Intervention): This will be treatment as usual without the patient decision aid

INTERVENTIONS:
Behavioral: Patient Decision Aid for Opioid Use Disorder — This will include information structured for patients about buprenorphine as a treatment options in the emergency department.
  Arms: Patient Decision Aid

SUMMARY:
This study aims to develop and pilot test a patient decision aid (PtDA) for emergency department (ED)-initiated buprenorphine treatment for opioid use disorder (OUD). The PtDA will be evaluated for acceptability, impact on patient knowledge, decisional conflict, and buprenorphine uptake compared to treatment as usual (TAU).

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18
* DSM-5 criteria for moderate-to-severe OUD
* Speaks and reads English
* Not currently prescribed MOUD
* Post-ED discharge patients with access to video/email

Exclusion Criteria:

- Prisoners

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2026-02-16 (Estimated); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Acceptability of Intervention Measure (AIM) | Day 1

SECONDARY OUTCOMES:
Knowledge about MOUD | pre and post intervention on day 1, and at 7 days
  This is a multiple choice knowledge quiz
Treatment selection | Day 1
Decisional Conflict Scale | Day 1
Receipt of buprenorphine | Day 1, 7

CONTACTS AND LOCATIONS:
Overall Officials: Lindsey Jennings, MD, MPH, Principal Investigator — Medical University of South Carolina
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified data will be shared via the NIDA data repository in accordance with NIH Data Management and Sharing Policy.
Supporting Information: Study Protocol